CLINICAL TRIAL: NCT02163057
Title: Prospective Study of HPV Specific Immunotherapy in Subjects With HPV Associated Head and Neck Squamous Cell Carcinoma (HNSCCa)
Brief Title: Study of HPV Specific Immunotherapy in Participants With HPV Associated Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPV-005
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Head and Neck Squamous Cell Cancer
Keywords: Head and neck squamous cell cancer; Papillomavirus
MeSH Terms: interventions — MEDI0457; VGX-3100; rocakinogene sifuplasmid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cohort 1: Surgery Cohort (Other): Participants received up to two doses of INO-3112 immunotherapy 3 weeks (± 3 days) apart before surgery and up to three doses of INO-3112 immunotherapy 3 weeks (± 3 days) apart after surgery for a total of no more than four doses of INO-3112 immunotherapy delivered IM followed by EP with CELLECTRA™-5P device.
  Interventions: Biological: INO-3112; Device: CELLECTRA™-5P
- Cohort 2: Chemoradiation (Other): Participants received four doses of INO-3112 immunotherapy delivered IM followed by EP with CELLECTRA™-5P device 3 weeks (± 3 days) apart beginning approximately 2 to 6 months after chemoradiation therapy.
  Interventions: Biological: INO-3112; Device: CELLECTRA™-5P

INTERVENTIONS:
Biological: INO-3112 — 1.1 mL of INO-3112 (VGX-3100 + INO-9012) delivered intramuscularly (IM) followed immediately by electroporation (EP) with CELLECTRA™-5P device for a total of 4 doses of immunotherapy.
  Other Names: VGX-3100; INO-9012
Device: CELLECTRA™-5P — CELLECTRA™-5P device was used for EP following IM delivery of INO-3112 for a total of 4 doses of immunotherapy.

SUMMARY:
This is a Phase I/IIa, open-label study to evaluate the safety, tolerability, and immunogenicity of INO-3112 DNA vaccine delivered by electroporation (EP) to participants with human papilloma virus (HPV) associated head and neck squamous cell cancer (HNSCC).

DETAILED DESCRIPTION:
This is a Phase I/IIa, open-label, study to evaluate the safety, tolerability, and immunogenicity of INO-3112 [6 mg of VGX-3100 (2 separate DNA plasmids respectively encoding E6 and E7 proteins of HPV 16 and HPV 18) and 1 mg of INO-9012 (DNA plasmid encoding human interleukin 12)] delivered by electroporation (EP) in up to 25 (twenty-five) participants with HPV positive head and neck cancer. The immunotherapy was studied in the following two groups of participants:

1. Participants who received immunotherapy before and after definitive surgery (Cohort I)
2. Participants who received immunotherapy at least 2 months after chemoradiation therapy (Cohort II).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written Ethics Committee approved informed consent.
2. Age ≥18 years.
3. Histologically confirmed HPV-positive (as assessed by p16 IHC or oncogenic HPV ISH or PCR) mucosal squamous cell head and neck cancer:

   * For pre-surgical participants, p16 positivity must be confirmed prior to the first dose.
   * For participants post-chemoradiation, HPV 16 and HPV 18 positivity must be confirmed prior to the first dose.
4. Adequate bone marrow, hepatic, and renal function. ANC (Absolute Neutrophil Count) ≥ 1.5x109 cell/ml, platelets ≥75,000 cells/mm3, hemoglobin ≥9.0 g/dL, concentrations of total serum bilirubin within 1.5 x upper limit of normal (ULN), (Aspartate Aminotransferase) AST, (Alanine Aminotransferase) ALT within 2.5x institutional ULN, (Creatine Phosphokinase) CPK within 2.5 x ULN.
5. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1.

Exclusion Criteria:

1. Anticipated concomitant immunosuppressive therapy (excluding non-systemic inhaled, topical skin and/or eye drop-containing corticosteroids).
2. Any concurrent condition requiring the continued use of systemic steroids (>10 mg prednisone or equivalent per day) or the use of immunosuppressive agents. All other corticosteroids must be discontinued at least 4 weeks prior to Day 0 of treatment.
3. Administration of any vaccine within 6 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Bagarazzi ML, Yan J, Morrow MP, Shen X, Parker RL, Lee JC, Giffear M, Pankhong P, Khan AS, Broderick KE, Knott C, Lin F, Boyer JD, Draghia-Akli R, White CJ, Kim JJ, Weiner DB, Sardesai NY. Immunotherapy against HPV16/18 generates potent TH1 and cytotoxic cellular immune responses. Sci Transl Med. 2012 Oct 10;4(155):155ra138. doi: 10.1126/scitranslmed.3004414. PMID 23052295
- [Background] Diehl MC, Lee JC, Daniels SE, Tebas P, Khan AS, Giffear M, Sardesai NY, Bagarazzi ML. Tolerability of intramuscular and intradermal delivery by CELLECTRA((R)) adaptive constant current electroporation device in healthy volunteers. Hum Vaccin Immunother. 2013 Oct;9(10):2246-52. doi: 10.4161/hv.24702. Epub 2013 Jun 4. PMID 24051434
- See also: Sponsor's Website — http://www.inovio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of HPV associated head and neck squamous cell carcinoma were enrolled in the study between 13th August 2014 to 23rd January 2017.
Period: Overall Study
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation
Started | 6 | 16
Completed | 3 | 11
Not Completed | 3 | 5
Not completed — Participant Refusal to Continue | 2 | 2
Not completed — Participant Significant Noncompliance | 0 | 1
Not completed — Progression of Disease | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study treatment plus EP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation | Total
Number analyzed (Participants) | 6 | 16 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (4.26) | 55.4 (10.26) | 57.3 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 6 | 14 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 16 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 5 | 14 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Event (SAEs)
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body, or worsening of a pre-existing condition, temporally associated with the use of a product whether or not considered related to the use of the product. TEAE is defined as any AE with onset after the administration of study medication through the end-of-study follow-up, or any event that was present at baseline but worsened in intensity or was subsequently considered treatment-related by the Investigator through the end of the study. Serious adverse event (SAE) is defined as an event that meets 1 of the following criteria: is fatal or life-threatening, results in persistent or significant disability or incapacity, constitutes a congenital anomaly or birth defect, is clinically meaningful or requires inpatient hospitalization or prolongation of existing hospitalization.
Time Frame: Up to 6 months post last dose
Population: Safety population included all participants who received at least one dose of study treatment plus EP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation
Number analyzed (Participants) | 6 | 16
Participants
  At least 1 TEAE | 6 | 15
  At least 1 Treatment-emergent SAE | 2 | 0

2. Secondary Outcome: E6 Antigen Specific Anti-HPV-16/18 Antibody Titers Assessed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Titers for HPV-16 and HPV-18 E6- and E7-specific antibodies were assessed by ELISA.
Time Frame: Up to 6 months post last dose
Population: Assigned Number of Doses (ANoD) population included all participants who received their assigned number of doses of study treatment plus EP. Number analyzed is the number of participants with data available for analysis at a specified time-point.
Measure: Mean (Standard Deviation); unit: log titer
Groups:
- Cohort 1: Surgery Cohort: Participants received up to two doses of INO-3112 immunotherapy 3 weeks (± 3 days) apart before surgery and up to three doses of INO-3112 immunotherapy 3 weeks (± 3 days) apart after surgery for a total of no more than four doses of INO-3112 immunotherapy delivered IM followed by EP with CELLECTRA™ device.
- Cohort 2: Chemoradiation: Participants received four doses of INO-3112 immunotherapy delivered IM followed by EP with CELLECTRA™ device 3 weeks (± 3 days) apart beginning approximately 2 to 6 months after chemoradiation therapy.
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation
Number analyzed (Participants) | 5 | 15
log titer
  HPV-16 ELISA titer, 1st dose: number analyzed (Participants) | 4 | 11
  HPV-16 ELISA titer, 1st dose | 3.6 (4.53) | 0.4 (1.18)
  HPV-16 ELISA titer, 2nd dose: number analyzed (Participants) | 4 | 13
  HPV-16 ELISA titer, 2nd dose | 2.2 (2.61) | 0.0 (0.00)
  HPV-16 ELISA titer, 3rd dose: number analyzed (Participants) | 5 | 13
  HPV-16 ELISA titer, 3rd dose | 2.6 (2.39) | 1.2 (2.33)
  HPV-16 ELISA titer, 4th dose: number analyzed (Participants) | 5 | 12
  HPV-16 ELISA titer, 4th dose | 2.4 (3.44) | 1.0 (2.42)
  HPV-16 ELISA titer, Week 2 post last dose: number analyzed (Participants) | 4 | 12
  HPV-16 ELISA titer, Week 2 post last dose | 2.8 (3.48) | 2.3 (2.91)
  HPV-16 ELISA titer, 1st long term follow-up: number analyzed (Participants) | 4 | 12
  HPV-16 ELISA titer, 1st long term follow-up | 1.3 (2.51) | 1.0 (2.42)
  HPV-16 ELISA titer, 2nd long term follow-up: number analyzed (Participants) | 5 | 10
  HPV-16 ELISA titer, 2nd long term follow-up | 0.0 (0.00) | 1.2 (2.63)
  HPV-16 ELISA titer, 3rd long term follow-up: number analyzed (Participants) | 2 | 9
  HPV-16 ELISA titer, 3rd long term follow-up | 0.0 (0.00) | 0.8 (2.40)
  HPV-16 ELISA titer, 4th long term follow-up: number analyzed (Participants) | 2 | 6
  HPV-16 ELISA titer, 4th long term follow-up | 0.0 (0.00) | 1.4 (3.39)
  HPV-16 ELISA titer, 5th long term follow-up: number analyzed (Participants) | 2 | 3
  HPV-16 ELISA titer, 5th long term follow-up | 0.0 (0.00) | 0.0 (0.00)
  HPV-16 ELISA titer, 6th long term follow-up: number analyzed (Participants) | 0 | 2
  HPV-16 ELISA titer, 6th long term follow-up |  | 3.1 (4.32)
  HPV-16 ELISA titer, initial surgery: number analyzed (Participants) | 5 | 0
  HPV-16 ELISA titer, initial surgery | 1.0 (2.24) |
  HPV-16 ELISA titer, surgery: number analyzed (Participants) | 4 | 0
  HPV-16 ELISA titer, surgery | 0.0 (0.00) |
  HPV-16 ELISA titer, follow-up Week 2 post-surgery: number analyzed (Participants) | 3 | 0
  HPV-16 ELISA titer, follow-up Week 2 post-surgery | 4.6 (1.27) |
  HPV-16 ELISA titer, optional surgery: number analyzed (Participants) | 1 | 0
  HPV-16 ELISA titer, optional surgery | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. |
  HPV-16 ELISA titer, unscheduled visit: number analyzed (Participants) | 1 | 0
  HPV-16 ELISA titer, unscheduled visit | 3.9 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. |
  HPV-16 ELISA titer, end of study follow-up: number analyzed (Participants) | 4 | 12
  HPV-16 ELISA titer, end of study follow-up | 0.0 (0.00) | 0.0 (0.00)
  HPV-18 ELISA titer, 1st dose: number analyzed (Participants) | 4 | 11
  HPV-18 ELISA titer, 1st dose | 0.0 (0.00) | 0.4 (1.18)
  HPV-18 ELISA titer, 2nd dose: number analyzed (Participants) | 4 | 13
  HPV-18 ELISA titer, 2nd dose | 0.0 (0.00) | 0.7 (1.69)
  HPV-18 ELISA titer, 3rd dose: number analyzed (Participants) | 5 | 13
  HPV-18 ELISA titer, 3rd dose | 0.0 (0.00) | 0.8 (1.88)
  HPV-18 ELISA titer, 4th dose: number analyzed (Participants) | 5 | 12
  HPV-18 ELISA titer, 4th dose | 1.0 (2.24) | 1.2 (2.12)
  HPV-18 ELISA titer, Week 2 post last dose: number analyzed (Participants) | 4 | 12
  HPV-18 ELISA titer, Week 2 post last dose | 0.0 (0.00) | 3.0 (3.25)
  HPV-18 ELISA titer, 1st long term follow-up: number analyzed (Participants) | 4 | 12
  HPV-18 ELISA titer, 1st long term follow-up | 1.3 (2.51) | 2.0 (3.04)
  HPV-18 ELISA titer, 2nd long term follow-up: number analyzed (Participants) | 5 | 10
  HPV-18 ELISA titer, 2nd long term follow-up | 1.0 (2.24) | 1.3 (2.09)
  HPV-18 ELISA titer, 3rd long term follow-up: number analyzed (Participants) | 2 | 9
  HPV-18 ELISA titer, 3rd long term follow-up | 0.0 (0.00) | 1.1 (2.28)
  HPV-18 ELISA titer, 4th long term follow-up: number analyzed (Participants) | 2 | 6
  HPV-18 ELISA titer, 4th long term follow-up | 0.0 (0.00) | 1.7 (2.68)
  HPV-18 ELISA titer, 5th long term follow-up: number analyzed (Participants) | 2 | 3
  HPV-18 ELISA titer, 5th long term follow-up | 0.0 (0.00) | 1.7 (2.89)
  HPV-18 ELISA titer, 6th long term follow-up: number analyzed (Participants) | 0 | 2
  HPV-18 ELISA titer, 6th long term follow-up |  | 6.1 (0.00)
  HPV-18 ELISA titer, initial surgery: number analyzed (Participants) | 5 | 0
  HPV-18 ELISA titer, initial surgery | 0.0 (0.00) |
  HPV-18 ELISA titer, surgery: number analyzed (Participants) | 4 | 0
  HPV-18 ELISA titer, surgery | 0.0 (0.00) |
  HPV-18 ELISA titer, follow-up Week 2 post-surgery: number analyzed (Participants) | 3 | 0
  HPV-18 ELISA titer, follow-up Week 2 post-surgery | 0.0 (0.00) |
  HPV-18 ELISA titer, optional surgery: number analyzed (Participants) | 1 | 0
  HPV-18 ELISA titer, optional surgery | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. |
  HPV-18 ELISA titer, unscheduled visit: number analyzed (Participants) | 1 | 0
  HPV-18 ELISA titer, unscheduled visit | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. |
  HPV-18 ELISA titer, end of study follow-up: number analyzed (Participants) | 4 | 12
  HPV-18 ELISA titer, end of study follow-up | 1.5 (3.05) | 2.8 (3.01)

3. Secondary Outcome: E7 Antigen Specific Anti-HPV-16/18 Antibody Titers Assessed by ELISA
Description: Titers for HPV-16 and HPV-18 E6- and E7-specific antibodies were assessed by ELISA.
Time Frame: Up to 6 months post last dose
Population: ANoD population included all participants who received their assigned number of doses of study treatment plus EP. Number analyzed is the number of participants with data available for analysis at a specified time-point.
Measure: Mean (Standard Deviation); unit: log titer
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation
Number analyzed (Participants) | 5 | 15
log titer
  HPV-16, 1st dose: number analyzed (Participants) | 4 | 11
  HPV-16, 1st dose | 0.0 (0.00) | 0.4 (1.18)
  HPV-16 ELISA titer, 2nd dose: number analyzed (Participants) | 4 | 13
  HPV-16 ELISA titer, 2nd dose | 0.0 (0.00) | 0.5 (1.69)
  HPV-16 ELISA titer, 3rd dose: number analyzed (Participants) | 5 | 13
  HPV-16 ELISA titer, 3rd dose | 1.2 (2.73) | 2.1 (2.85)
  HPV-16 ELISA titer, 4th dose: number analyzed (Participants) | 5 | 12
  HPV-16 ELISA titer, 4th dose | 3.0 (3.06) | 3.0 (3.41)
  HPV-16 ELISA titer, Week 2 post last dose: number analyzed (Participants) | 4 | 12
  HPV-16 ELISA titer, Week 2 post last dose | 2.8 (3.48) | 3.3 (4.09)
  HPV-16 ELISA titer, 1st long term follow-up: number analyzed (Participants) | 4 | 12
  HPV-16 ELISA titer, 1st long term follow-up | 2.5 (3.03) | 2.8 (3.63)
  HPV-16 ELISA titer, 2nd long term follow-up: number analyzed (Participants) | 5 | 10
  HPV-16 ELISA titer, 2nd long term follow-up | 0.8 (1.75) | 1.6 (3.28)
  HPV-16 ELISA titer, 3rd long term follow-up: number analyzed (Participants) | 2 | 9
  HPV-16 ELISA titer, 3rd long term follow-up | 0.0 (0.00) | 1.5 (3.24)
  HPV-16 ELISA titer, 4th long term follow-up: number analyzed (Participants) | 2 | 6
  HPV-16 ELISA titer, 4th long term follow-up | 0.0 (0.00) | 0.8 (2.05)
  HPV-16 ELISA titer, 5th long term follow-up: number analyzed (Participants) | 2 | 3
  HPV-16 ELISA titer, 5th long term follow-up | 0.0 (0.00) | 3.1 (5.43)
  HPV-16 ELISA titer, 6th long term follow-up: number analyzed (Participants) | 0 | 2
  HPV-16 ELISA titer, 6th long term follow-up |  | 4.2 (5.87)
  HPV-16 ELISA titer, initial surgery: number analyzed (Participants) | 5 | 0
  HPV-16 ELISA titer, initial surgery | 0.0 (0.00) |
  HPV-16 ELISA titer, surgery: number analyzed (Participants) | 4 | 0
  HPV-16 ELISA titer, surgery | 0.0 (0.00) |
  HPV-16 ELISA titer, follow-up Week 2 post-surgery: number analyzed (Participants) | 3 | 0
  HPV-16 ELISA titer, follow-up Week 2 post-surgery | 0.0 (0.00) |
  HPV-16 ELISA titer, optional surgery: number analyzed (Participants) | 1 | 0
  HPV-16 ELISA titer, optional surgery | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. |
  HPV-16 ELISA titer, unscheduled visit: number analyzed (Participants) | 1 | 0
  HPV-16 ELISA titer, unscheduled visit | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. |
  HPV-16 ELISA titer, end of study follow-up: number analyzed (Participants) | 4 | 12
  HPV-16 ELISA titer, end of study follow-up | 0.0 (0.00) | 1.3 (2.45)
  HPV-18 ELISA titer, 1st dose: number analyzed (Participants) | 4 | 11
  HPV-18 ELISA titer, 1st dose | 0.0 (0.00) | 0.5 (1.51)
  HPV-18 ELISA titer, 2nd dose: number analyzed (Participants) | 4 | 13
  HPV-18 ELISA titer, 2nd dose | 2.5 (2.89) | 0.3 (1.08)
  HPV-18 ELISA titer, 3rd dose: number analyzed (Participants) | 5 | 13
  HPV-18 ELISA titer, 3rd dose | 2.7 (3.67) | 1.3 (2.03)
  HPV-18 ELISA titer, 4th dose: number analyzed (Participants) | 5 | 12
  HPV-18 ELISA titer, 4th dose | 4.5 (4.17) | 3.0 (3.21)
  HPV-18 ELISA titer, Week 2 post last dose: number analyzed (Participants) | 4 | 12
  HPV-18 ELISA titer, Week 2 post last dose | 8.0 (1.65) | 4.2 (2.83)
  HPV-18 ELISA titer, 1st long term follow-up: number analyzed (Participants) | 4 | 12
  HPV-18 ELISA titer, 1st long term follow-up | 6.9 (2.44) | 4.5 (3.41)
  HPV-18 ELISA titer, 2nd long term follow-up: number analyzed (Participants) | 5 | 10
  HPV-18 ELISA titer, 2nd long term follow-up | 5.8 (3.98) | 1.8 (3.13)
  HPV-18 ELISA titer, 3rd long term follow-up: number analyzed (Participants) | 2 | 9
  HPV-18 ELISA titer, 3rd long term follow-up | 2.0 (2.77) | 3.1 (3.79)
  HPV-18 ELISA titer, 4th long term follow-up: number analyzed (Participants) | 2 | 6
  HPV-18 ELISA titer, 4th long term follow-up | 0.0 (0.00) | 2.5 (2.83)
  HPV-18 ELISA titer, 5th long term follow-up: number analyzed (Participants) | 2 | 3
  HPV-18 ELISA titer, 5th long term follow-up | 0.0 (0.00) | 5.5 (4.80)
  HPV-18 ELISA titer, 6th long term follow-up: number analyzed (Participants) | 0 | 2
  HPV-18 ELISA titer, 6th long term follow-up |  | 8.3 (0.00)
  HPV-18 ELISA titer, initial surgery: number analyzed (Participants) | 5 | 0
  HPV-18 ELISA titer, initial surgery | 0.0 (0.00) |
  HPV-18 ELISA titer, surgery: number analyzed (Participants) | 4 | 0
  HPV-18 ELISA titer, surgery | 2.4 (4.70) |
  HPV-18 ELISA titer, follow-up Week 2 post-surgery: number analyzed (Participants) | 3 | 0
  HPV-18 ELISA titer, follow-up Week 2 post-surgery | 1.3 (2.26) |
  HPV-18 ELISA titer, optional surgery: number analyzed (Participants) | 1 | 0
  HPV-18 ELISA titer, optional surgery | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. |
  HPV-18 ELISA titer, unscheduled visit: number analyzed (Participants) | 1 | 0
  HPV-18 ELISA titer, unscheduled visit | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. |
  HPV-18 ELISA titer, end of study follow-up: number analyzed (Participants) | 4 | 12
  HPV-18 ELISA titer, end of study follow-up | 4.4 (5.29) | 4.6 (3.03)

4. Secondary Outcome: Change From Baseline (CFB) in Combined HPV-16 and HPV-18 E6 and E7 Antigen-Specific Spot-Forming Units Per Million Peripheral Blood Mononuclear Cell (SFU/10^6 PBMC) as Assessed by Enzyme-Linked Immunosorbent Spot-Forming Assay (ELISpot)
Time Frame: Baseline up to 6 months post last dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SFU/10^6 PBMC
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation
Number analyzed (Participants) | 5 | 15
SFU/10^6 PBMC
  Baseline | 20.3 (22.65) | 11.7 (10.25)
  CFB at 2nd dose: number analyzed (Participants) | 4 | 13
  CFB at 2nd dose | 24.2 (34.56) | 96.9 (118.41)
  CFB at 3rd dose: number analyzed (Participants) | 4 | 15
  CFB at 3rd dose | 15.0 (17.54) | 158.9 (231.73)
  CFB at 4th dose: number analyzed (Participants) | 5 | 13
  CFB at 4th dose | 50.3 (49.06) | 263.6 (597.80)
  CFB at Week 2 post last dose: number analyzed (Participants) | 4 | 14
  CFB at Week 2 post last dose | 68.3 (63.98) | 354.7 (632.29)
  CFB at 1st long term follow-up: number analyzed (Participants) | 4 | 11
  CFB at 1st long term follow-up | 182.2 (211.31) | 128.8 (132.05)
  CFB at 2nd long term follow-up: number analyzed (Participants) | 5 | 7
  CFB at 2nd long term follow-up | 102.3 (140.03) | 151.1 (94.32)
  CFB at 3rd long term follow-up: number analyzed (Participants) | 2 | 7
  CFB at 3rd long term follow-up | 127.6 (3.46) | 113.2 (153.59)
  CFB at 4th long term follow-up: number analyzed (Participants) | 1 | 4
  CFB at 4th long term follow-up | 41.4 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. | 29.8 (28.11)
  CFB at 5th long term follow-up: number analyzed (Participants) | 2 | 1
  CFB at 5th long term follow-up | 129.1 (19.87) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  CFB at 6th long term follow-up: number analyzed (Participants) | 1 | 1
  CFB at 6th long term follow-up | 141.7 (NA) — Standard deviation could not be calculated due to an insufficient number of participants. | 11.7 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  CFB at follow-up Week 2 post-surgery: number analyzed (Participants) | 2 | 0
  CFB at follow-up Week 2 post-surgery | 154.2 (168.50) |
  CFB at end of study follow-up: number analyzed (Participants) | 4 | 9
  CFB at end of study follow-up | 50.0 (42.75) | 70.5 (87.09)

5. Secondary Outcome: Change From Baseline (CFB) in CD8+ T-Cell Responses Specific for HPV-16 as Assessed by Flow Cytometry
Description: A flow cytometry assay called "lytic granule loading" was used to analyze CD8+ T cells specific for HPV-16 and CD8+ T cells specific for HPV-18 by evaluating the following markers: CD8, granzyme A (GrzA), granzyme B (GrzB), and perforin (Prf) co-expression with CD137, CD69, or CD38.
Time Frame: At baseline and Week 2 post last dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells/million T-cells
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation
Number analyzed (Participants) | 5 | 15
cells/million T-cells
  CD8+CD137+GrzA+GrzB+Prf+, baseline: number analyzed (Participants) | 2 | 6
  CD8+CD137+GrzA+GrzB+Prf+, baseline | 0.09 (0.124) | 0.02 (0.039)
  CD8+CD137+GrzA+GrzB+Prf+,CFB Week 2 post last dose: number analyzed (Participants) | 2 | 6
  CD8+CD137+GrzA+GrzB+Prf+,CFB Week 2 post last dose | 0.16 (0.230) | 0.11 (0.188)
  CD8+CD69+GrzA+GrzB+Prf+, baseline: number analyzed (Participants) | 2 | 6
  CD8+CD69+GrzA+GrzB+Prf+, baseline | 0.00 (0.000) | 0.17 (0.345)
  CD8+CD69+GrzA+GrzB+Prf+, CFB Week 2 post last dose: number analyzed (Participants) | 2 | 6
  CD8+CD69+GrzA+GrzB+Prf+, CFB Week 2 post last dose | 0.48 (0.282) | 0.20 (0.471)
  CD8+CD38+GrzA+GrzB+Prf+, baseline: number analyzed (Participants) | 2 | 6
  CD8+CD38+GrzA+GrzB+Prf+, baseline | 0.00 (0.000) | 0.14 (0.163)
  CD8+CD38+GrzA+GrzB+Prf+, CFB Week 2 post last dose: number analyzed (Participants) | 2 | 6
  CD8+CD38+GrzA+GrzB+Prf+, CFB Week 2 post last dose | 0.89 (0.457) | 0.26 (0.555)

6. Secondary Outcome: Change From Baseline (CFB) in CD8+ T-Cell Responses Specific for HPV-18 as Assessed by Flow Cytometry
Description: as for outcome 5
Time Frame: At baseline and Week 2 post last dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells/million T-cells
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation
Number analyzed (Participants) | 5 | 15
cells/million T-cells
  CD8+CD137+GrzA+GrzB+Prf+, baseline: number analyzed (Participants) | 2 | 6
  CD8+CD137+GrzA+GrzB+Prf+, baseline | 0.00 (0.000) | 0.05 (0.070)
  CD8+CD137+GrzA+GrzB+Prf+,CFB Week 2 post last dose: number analyzed (Participants) | 2 | 6
  CD8+CD137+GrzA+GrzB+Prf+,CFB Week 2 post last dose | 0.09 (0.073) | 0.07 (0.089)
  CD8+CD69+GrzA+GrzB+Prf+, baseline: number analyzed (Participants) | 2 | 6
  CD8+CD69+GrzA+GrzB+Prf+, baseline | 0.00 (0.000) | 0.10 (0.158)
  CD8+CD69+GrzA+GrzB+Prf+, CFB Week 2 post last dose: number analyzed (Participants) | 2 | 6
  CD8+CD69+GrzA+GrzB+Prf+, CFB Week 2 post last dose | 0.20 (0.283) | 0.34 (0.540)
  CD8+CD38+GrzA+GrzB+Prf+, baseline: number analyzed (Participants) | 2 | 6
  CD8+CD38+GrzA+GrzB+Prf+, baseline | 0.00 (0.000) | 0.06 (0.135)
  CD8+CD38+GrzA+GrzB+Prf+, CFB Week 2 post last dose: number analyzed (Participants) | 2 | 6
  CD8+CD38+GrzA+GrzB+Prf+, CFB Week 2 post last dose | 0.73 (0.841) | 0.36 (0.552)

7. Secondary Outcome: Mean Difference in Tumor Infiltrating Lymphocytes (TILs) in Presurgical and Surgical Tumor Tissue Samples of Cohort I as Assessed by Immunohistochemistry (IHC)
Description: The difference in means (post-surgery minus screening) for tumor-infiltrating lymphocytes (TILs) such as CD8, FoxP3, and perforin was analyzed using immunohistochemistry staining techniques.
Time Frame: At screening and post-surgery
Population: ANoD population included all participants who received their assigned number of doses of study treatment plus EP.
Measure: Mean (95% Confidence Interval); unit: positive cells per square millimeter
Arm/Group | Cohort 1: Surgery Cohort
Number analyzed (Participants) | 4
positive cells per square millimeter
  CD8 | 268.5 [-1583.5 to 2120.5]
  FoxP3 | -79.8 [-834.2 to 674.7]
  Perforin | 9.5 [-0.4 to 19.4]

8. Secondary Outcome: Mean Difference in CD8/FoxP3 Ratio in Presurgical and Surgical Tumor Tissue Samples of Cohort I as Assessed by Immunohistochemistry (IHC)
Description: The difference in means (post-surgery minus screening) for the CD8/FoxP3 ratio was analyzed using immunohistochemistry staining techniques.
Time Frame: At screening and post-surgery
Population: ANoD population included all participants who received their assigned number of doses of study treatment plus EP.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: Surgery Cohort
Number analyzed (Participants) | 4
ratio | 0.2 [-0.8 to 1.2]

9. Secondary Outcome: Phenotype of Cultured TILs
Time Frame: Up to 6 months post last dose
Population: Data was not collected due to lack of recoverable samples sufficient for analysis
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months post last dose
Arm/Group | Cohort 1: Surgery Cohort | Cohort 2: Chemoradiation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/16
Other Adverse Events (participants affected / at risk) | 6/6 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Surgery Cohort (N=6) | Cohort 2: Chemoradiation (N=16)
Anaphylactic reaction (Immune system disorders) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Surgery Cohort (N=6) | Cohort 2: Chemoradiation (N=16)
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Thyroiditis (Endocrine disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 1
Eructation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 3
Glossodynia (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oral Discomfort (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1
Salivary Duct Inflammation (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Tongue Discolouration (Gastrointestinal disorders) | 1 | 0
Tongue Oedema (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Injection Site Bruising (General disorders) | 2 | 3
Injection Site Erythema (General disorders) | 2 | 5
Injection Site Induration (General disorders) | 0 | 1
Injection Site Pain (General disorders) | 5 | 10
Injection Site Swelling (General disorders) | 1 | 4
Localised Oedema (General disorders) | 2 | 0
Mucosal Inflammation (General disorders) | 1 | 1
Seasonal Allergy (Immune system disorders) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 2 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 2
Oral Herpes (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 2 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2
Neuropathy Peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1
Restless Legs Syndrome (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia Areata (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Fibrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Neoplasm Excision (Surgical and medical procedures) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT02163057/Prot_SAP_001.pdf